CLINICAL TRIAL: NCT03537833
Title: Association Between Proton Pump Inhibitors and the Incidence of Hematologic Toxicity of Pemetrexed: a Prospective, Multicenter, Observational and Longitudinal Study Among Patients Treated by a Pemetrexed-based Chemotherapy
Brief Title: Association Between Proton Pump Inhibitors and Hematologic Toxicity of Pemetrexed
Acronym: IPPEM
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18047*
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Patients With Non-small Cell Lung Cancer (NSCLC) and Pleural Mesothelioma and Treated With a Pemetrexed-based Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "PPI-positive" or "test group": Patients treated with PPI
  Interventions: Other: pemetrexed-related hematological toxicity
- "PPI-negative" or "control group": Patients not treated with PPI
  Interventions: Other: pemetrexed-related hematological toxicity

INTERVENTIONS:
Other: pemetrexed-related hematological toxicity — hematological toxicity will be found on biologic data the day or the day before chemotherapy. Classification will based on NCI-CTCAE criteria

SUMMARY:
Pemetrexed is a multi-folate inhibitor approved in the treatment of non-small cell lung cancer (NSCLC) and pleural mesothelioma. Its toxicity profile is mainly hematologic (anemia, neutropenia and thrombopenia) and can be limiting when > grade 2 according to NCI-CTCAE criteria. First clinical trials highlighted hematologic toxicity, especially anemia, which was reduced by decreasing pemetrexed dosage from 600 to 500 mg/m² Q3W and by adding systematic vitamin supplementation (B9/B12). Despite this, incidence of hematological toxicity remains frequent with anemia occurring in more than 20% of patients treated by pemetrexed in combination. Methotrexate, a well-known antineoplastic drugs used in several cancer and non-cancer disease conditions can also induced severe hematologic toxicity in case of methotrexate-reduced elimination and, as a consequence, its accumulation. For example, the elimination of methotrexate is mediated by tubular secretion through type 1 and type 3 organic anion transport (hOAT1 and hOAT3). Association with drugs that inhibits hOATs can induced a hematological toxicity caused by methotrexate accumulation. Among these, proton pump inhibitors (PPIs) are known to inhibit hOATs. The drug interaction that results from their combination with methotrexate is clinically relevant and lead to an increased hematological toxicity. However, hypothetical drug interaction between PPIs and pemetrexed is unknown while pemetrexed seems to be mostly eliminated by hOAT3 (11-fold higher than methotrexate). One study revealed lansoprazole to inhibits in vitro hOAT3. This same study investigates in a retrospective chart patients treated by pemetrexed and the study found a significant association between combination with PPI and hematological toxicity by pemetrexed. Unfortunately this study lacks of relevant methodology and suffered from its retrospective chart. This potential drug interaction must be a real concern for oncologists and clinical pharmacists. The investigators aim to investigate the potential association between PPIs and pemetrexed combination and the incidence of hematological toxicity in a multicenter and prospective study.

DETAILED DESCRIPTION:
Prospective, longitudinal, multicenter and observational study. All eligible patients will receive clear information about aims and research modalities on the medical consultation and before first course of chemotherapy. If patient agrees with study aims and protocol, disease and therapeutic management will not be change.

Research agree and participation leads to

Data collection:

* Clinical data: weight, height, body mass index

  1. Demographic data: sociodemographic data, comorbidities
  2. Disease data: related to tumor disease and antineoplastic protocol including adjuvant medications like antiemetic of antidiarrheal agents for example.
* complete medication review: a minimum of 3 information sources among the patient and/or family and close, patient health records, community pharmacy, general practitioner,
* activation of a specific study patient record
* biologic data collection: blood count and thrombocythemia during all period study and three week after patient study completion,
* supplementary data in case of hematologic toxicity: hospitalization, growth factors (like erythropoietin and/or granulocyte colony-stimulating factor use), blood transfusions, intravenous iron, chemotherapy treatment delay All patients are followed since inclusion and for 18 months. Research logistic Patients will be recruited in cancer hospital service where patients received pemetrexed in the four study participant centers. Full information and all necessary clarification about study will be explained to all eligible patients with an appropriate consent form. Data collection using case report form will be performed by pharmacists and physicians from hospitalization setting.

Recruiting duration period Twelve months

Subject duration period Eighteen months Subject accessibility Patients will be recruited in one of the four participant centers Statistical analysis Number of patients to include with statistical considerations

It is planned to include 100 patients per group after calculating the number of subjects required (nQuery software) taking into account the following assumptions:

* Risk alpha = 0.05
* Statistical power = 90%
* Percentage of patients without hematologic toxicity in PPI-negative group = 0.62
* Percentage of patients without hematologic toxicity in PPI-positive group = 0.88 (Hazard ratio = 3.74) Statistical analysis methods of criteria Data description will be performed using mean and standard deviation or median (interquartile interval and minimum and maximum) for quantitative variables according to variable distribution and number and percentage for qualitative variables.

Bivariate analysis will be conducted in order to found the association between hematological toxicity or not and clinical variables. Multivariate analysis will be performed with Cox model, using a dependent variable "presence or not of a hematologic toxicity" and independents variables, variables that are associated with a "p" less than 0.20 with confusion factors adjustment.

Treatment of missing data The study will be performed in order to minimize the number of missing data. For each variable number and percentage of missing data will be described.

ELIGIBILITY:
Inclusion criteria :

* Patients who receive a pemetrexed-based chemotherapy regimen for the treatment of non-small cell lung cancer (NSCLC) or mesothelioma,
* Patients who consent to participate,
* Patients for whom it is possible to characterize the consumption of proton pump inhibitors with name of the PPI and dosage.

Exclusion criteria :

* Patients who receive pemetrexed out of intravenous of for another condition than NSCLC or mesothelioma
* Patients under 18 or who refused the participation in the data collection,
* Patient previously treated by a pemetrexed-based chemotherapy,
* Patients who first receive a pemetrexed-based regimen with an initial dose adjustment (<500 mg/m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive a pemetrexed-based chemotherapy regimen for the treatment of non-small cell lung cancer (NSCLC) or mesothelioma
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Association between PPI consumption and pemetrexed-related hematological toxicity (grade ≥ 3) | Day 0
  The hematological toxicity will be found on biologic data the day or the day before chemotherapy. Classification will based on NCI-CTCAE criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Slimano F, Le Bozec A, Cransac A, Foucher P, Lesauvage F, Delclaux B, Dory A, Mennecier B, Bertrand B, Gubeno-Dumon MC, Dukic S, Mongaret C, Bouche O, Hettler D, Boulin M, Dewolf M, Kanagaratnam L. Association between proton pump inhibitors and severe hematological toxicity in patients receiving pemetrexed-based anticancer treatment: The prospective IPPEM study. Lung Cancer. 2022 Apr;166:114-121. doi: 10.1016/j.lungcan.2022.02.007. Epub 2022 Feb 24. PMID 35263663